CLINICAL TRIAL: NCT03411694
Title: Patient Perception on the Role of Anesthesiologists: a Survey on the Belgian Perspective
Brief Title: Patient Perception on the Role of Anesthesiologists
Status: Completed | Type: Observational
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Stessel Björn, Principal Investigator, Anesthesiologist, MD, PhD, Jessa Hospital
Other Study IDs: 18.04/anesth18.01
Record Dates: First submitted 2018-01-11; First posted 2018-01-26 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Anesthesia; Surgery
Keywords: Survey; Anesthesia; Anesthesiologist; Patient perspective
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Survey in patients from the Jessa Hospital that are planned for elective surgery, both ambulatory and inpatient.

SUMMARY:
Previous studies showed that the role of the anesthesiologist, their education and role within the hospital is not known by the general public. The lack of knowledge about anesthesia can be an important factor in patients' fear before the planned surgery and can therefore impact patient's general satisfaction. By means of a survey in patients planned for elective surgery, the investigators want to investigate the perception of patients regarding the anesthesiologist, their education and role within the hospital, the general knowledge of the patient regarding anesthesia and possible pre-operative fears and concerns.

DETAILED DESCRIPTION:
Introduction:

Previous studies, mainly performed in the USA and a few in Europe, showed that the role of the anesthesiologist, their education and role within the hospital is not known by the general public (1). Other studies questioned the expectations as well as fear of patients with respect to anesthesia (2). The lack of knowledge about the anesthesia can be an important factor in patients' fear before the planned surgery and can therefore impact patient's general satisfaction. While studies have been performed in several countries, not a single study as far as the investigators know, has been performed in Belgium. Given the fact that the anesthesiologist plays an important role during all stages of surgery (pre-, per-, post-operative), it is important to know how patients experience anesthesia and the role of the anesthesiologist. In this way, possible points of attention can be explored which can lead to a better patient satisfaction in the future.

Outcome measures:

With this study, the investigators want to investigate the perception of patients regarding the anesthesiologist, their education and role within the hospital, the general knowledge of the patient regarding anesthesia and possible pre-operative fears and concerns.

The investigators will determine these outcome measures by performing a survey (standardized questions) which will investigate the following 8 parts:

* Patient demographics
* The perception of the role and educational training of the anesthesiologist
* The role of the anesthesiologist in the hospital
* General knowledge of anesthesia
* Trust in medical specialist and anesthesiologist
* Fear and concerns about anesthesia
* Patients' expectation regarding recovery and postoperative pain
* Information for the anesthesiologist and possible points of improvement

Design:

In this monocentric, investigator-initiated, observational, cohort-study, the investigators will perform a survey in all patients that are planned to undergo elective surgery, both ambulatory as well as inpatient surgery. This study will be performed according to the Declaration of Helsinki and will be approved by the Ethical Committee of the Jessa Hospital before the start of the study. A written informed consent will be obtained before participation in the study.

Study Procedures:

Patients that are planned for elective surgery, both ambulatory and inpatient surgery, will be contacted by a researcher prior to the surgery and asked to participate in the study. After a written informed consent is obtained, the survey will be performed by a single researcher, to minimize inter-individual variability. During the survey, family or other people present in the hospital room are not allowed to help the patient. In hospital rooms where more than 1 patient is present, the survey will be performed only once.

Statistical analysis:

Based on previous, comparable studies (1,3,4), 350 patients will be included in this study. Descriptive statistics will be presented as frequencies and percentages of the total amount of patients for categorical variables, while numerical variables will be presented as mean ± SD. Multiple linear regression analysis and correlations will be calculated (depending on normality). A p-value <0.05 is considered statistical significant, while p<0.10 is considered a tendency.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of age
* American Society of Anesthesiology (ASA) physical status classification: 1-3
* Patients planned to undergo surgery (both ambulatory and inpatient surgery)
* Patients that speak Dutch, French or English

Exclusion Criteria:

* Patients that don't speak Dutch, French or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients from the Jessa Hospital, that are planned for elective surgery (both ambulatory and inpatient surgery)
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
The role and educational training of the anesthesiologist | max 1 hour per survey
  The patients' perception of the work and educational training of the anesthesiologist

SECONDARY OUTCOMES:
Patient demographics | max 1 hour per survey
  Gender, age, highest education level, nationality, language, medical condition
The role of the anesthesiologist in the hospital | max 1 hour per survey
  The patients' perception of the workplace of an anesthesiologist in the hospital
General knowledge of anesthesia | max 1 hour per survey
  The patients' perception of anesthesia in general
Trust in medical specialist and anesthesiologist | max 1 hour per survey
  The patients' trust in the medical specialist and anesthesiologist
Fear and concerns about anesthesia | max 1 hour per survey
  The patients' fear and concerns before the surgery
Recovery and postoperative pain | max 1 hour per survey
  Several questions regarding the patients' expectation of recovery and postoperative pain
Information for the anesthesiologist and possible points of improvement | max 1 hour per survey
  Possible points of improvement for the anesthesiologist

CONTACTS AND LOCATIONS:
Overall Officials: Björn Stessel, MD, PhD, Principal Investigator — Jessa Hospital, Dep. of Anesthesiology
Locations (1):
- Jessa Hospital, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nagrampa D, Bazargan-Hejazi S, Neelakanta G, Mojtahedzadeh M, Law A, Miller M. A survey of anesthesiologists' role, trust in anesthesiologists, and knowledge and fears about anesthesia among predominantly Hispanic patients from an inner-city county preoperative anesthesia clinic. J Clin Anesth. 2015 Mar;27(2):97-104. doi: 10.1016/j.jclinane.2014.05.012. Epub 2015 Jan 17. PMID 25605048
- [Background] Chew ST, Tan T, Tan SS, Ip-Yam PC. A survey of patients' knowledge of anaesthesia and perioperative care. Singapore Med J. 1998 Sep;39(9):399-402. PMID 9885718
- [Background] Hariharan S, Merritt-Charles L, Chen D. Patient perception of the role of anesthesiologists: a perspective from the Caribbean. J Clin Anesth. 2006 Nov;18(7):504-9. doi: 10.1016/j.jclinane.2006.03.004. PMID 17126778
- [Background] Gottschalk A, Seelen S, Tivey S, Gottschalk A, Rich G. What do patients know about anesthesiologists? Results of a comparative survey in an U.S., Australian, and German university hospital. J Clin Anesth. 2013 Mar;25(2):85-91. doi: 10.1016/j.jclinane.2012.06.017. Epub 2013 Jan 17. PMID 23333789